CLINICAL TRIAL: NCT06817434
Title: Study on Evaluating the Effectiveness of Statins in the Treatment of Moyamoya Disease
Acronym: SEST-MOYA
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023-297-02
Record Dates: First submitted 2025-01-26; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Revascularization/Conservative management — Revascularization/Conservative management

SUMMARY:
The purpose of this study is to investigate the effectiveness of statins in the treatment of moyamoya disease based on multimodal magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

1. The imaging examination meets the diagnostic criteria for moyamoya disease;
2. Sign the informed consent form;
3. Age ≥18 years old;
4. Baseline mRS score ≤2 points;
5. The patient receives revascularization/conservative treatment;
6. There is at least 1 imaging follow-up result.

Exclusion Criteria:

1. Patients with atherosclerosis, autoimmune diseases, meningitis, Down syndrome, cranial trauma, or those who have undergone radioactive head irradiation, as these conditions may lead to secondary cerebrovascular disease and contribute to the development of Moyamoya syndrome;
2. Individuals under the age of 18;
3. Participants who refuse to take part in this study;
4. Pregnant patients;
5. Those with concurrent intracranial aneurysms, cerebrovascular malformations, brain tumors, or hydrocephalus;
6. A history of stroke occurring more than three months prior to the diagnosis of Moyamoya disease;
7. Individuals with a history of coronary heart disease or previous cardiovascular and cerebrovascular surgical interventions, including cerebral revascularization, intracranial artery stent implantation, carotid artery stenting, endarterectomy, coronary artery bypass grafting, or coronary stent implantation;
8. Allergies to contrast media;
9. Patients with missing imaging data or whose image quality cannot be analyzed;
10. Individuals who refuse or are unable to undergo imaging follow-up;
11. Patients receiving other types of lipid-lowering drug treatments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with MMD in Beijing Tiantan Hospital will be recruited. Eligibility will be determined through a checklist of inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participants experiencing cerebrovascular events (TIA, ischemic stroke, or hemorrhagic stroke) | 18 months during follow-up
  The occurrence of cerebrovascular events, including TIA, ischemic stroke, or hemorrhagic stroke, will be assessed over an 18-month follow-up period.

SECONDARY OUTCOMES:
Changes in Neurological Function (mRS, NIHSS) at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  The mRS and NIHSS will be used to assess changes in neurological function at 12 and 18 months after treatment.
Changes in Cognitive Function (MoCA, MMSE) at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  The MoCA and MMSE will be used to evaluate changes in cognitive function at 12 and 18 months after treatment.
Structural Remodeling of the Internal Carotid Artery Terminal and Middle Cerebral Artery Wall at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  High-resolution magnetic resonance vessel wall imaging will be used to evaluate structural remodeling changes in the internal carotid artery terminal and middle cerebral artery wall at 12 and 18 months after treatment.
Changes in Cerebral Blood Perfusion at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  ASL will be used to assess cerebral blood perfusion changes at 12 and 18 months after treatment.
Rate of New Cerebral Infarcts at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  The occurrence of new cerebral infarcts at 12 and 18 Months after treatment will be evaluated using MRI.
Hemodynamic Changes at the Internal Carotid Artery Terminal at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  4D-Flow MRI and hemodynamic analysis will be used to evaluate changes in hemodynamics at the internal carotid artery terminal at 12 and 18 months after treatment.
Changes in Blood Lipid Levels at 12 and 18 Months After Treatment | 12 and 18 months during follow-up
  Blood lipid levels will be measured and compared at 12 and 18 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China, China